CLINICAL TRIAL: NCT01447121
Title: Tatsu/Tradewind System User Performance Evaluation
Brief Title: User Study of an Investigational Blood Glucose Monitoring System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ascensia Diabetes Care (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CTD-PRO-2011-005-01
Record Dates: First submitted 2011-10-04; First posted 2011-10-06 (Estimated); Results first posted 2012-10-22 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-01

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intended Users of the System (Experimental): Untrained subjects with diabetes use an investigational blood glucose monitoring system (Tatsu/Tradewind Investigational BG Monitoring System) to self-test capillary blood obtained from fingerstick.
  Interventions: Device: Tatsu/Tradewind Investigational BG Monitoring System

INTERVENTIONS:
Device: Tatsu/Tradewind Investigational BG Monitoring System — Tradewind is a Bayer investigational meter that used an investigational sensor.

SUMMARY:
This clinical trial is designed to assess an investigational blood glucose monitoring system with fingerstick blood in the hands of untrained intended users.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or type 2 diabetes
* 18 years of age and older
* Able to speak, read, and understand English
* Willing to complete all study procedures

Exclusion Criteria:

* Previously participated in a study using this investigational system
* Working for a medical laboratory, hospital, or other clinical setting that involves training on and clinical use of blood glucose monitors
* Pregnancy
* Hemophilia or any other bleeding disorder
* Working for a competitive medical device company or having an immediate family member or someone who is not a family member but is living within the household of someone who works for such a company
* A condition which, in the opinion of the investigator, would put the person or study conduct at risk (reason for exclusion will be clearly documented by investigator or designee).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2011-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Bailey, MD, Principal Investigator — AMCR Institute
Locations (1):
- AMCR Institute, Escondido, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Intended Users of the System: Untrained subjects with diabetes use an investigational blood glucose monitoring system (Tatsu/Tradewind Investigational BG Monitoring System) to self-test capillary blood obtained from fingerstick.
  Tatsu/Tradewind Investigational BG Monitoring System : Tradewind is a Bayer investigational meter that used an investigational sensor.
Period: Overall Study
Arm/Group | Intended Users of the System
Started | 118
Completed | 118
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Intended Users of the System: Study results from 2 subjects were excluded from all data analysis, because study staff inadvertently performed study tasks that could be considered 'training' them. (According to protocol, training was not allowed.)
Arm/Group | Intended Users of the System
Number analyzed (Participants) | 116
Age, Customized [Mean (Full Range); unit: years] | 52.3 [18 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61
  Male | 55
Region of Enrollment [Number; unit: participants]
  United States | 116

OUTCOME MEASURES:

1. Primary Outcome: Number of Self-Test Fingerstick Blood Glucose (BG) Results Within +/- 15mg/dL (<75 mg/dL) or Within +/- 20% (>=75 mg/dL) of Laboratory Glucose Method
Description: Untrained subjects with diabetes tested self-test fingerstick blood using an investigational Blood Glucose Monitoring System (BGMS), which included an investigational meter and sensor. BGM results were compared with capillary plasm BG results obtained with a reference lab glucose method - Yellow Springs Instrument (YSI) Analyzer. BG meter results were used to calculate the number of BG results within +/- 15 mg/dL (for reference BG results <75mg/dL) or +/- 20% (for reference BG results >=75mg/dL) of the reference method results (YSI capillary plasma).
Time Frame: 1 hour
Population: 115(115x1)test results are possible. 118 subjects tested one of 3 test strip lots on the BGM system. Study results from 2 subjects were excluded from all data analyses as already described. One subject test exceeded time interval (defined in protocol) between meter test and reference method.
Measure: Number; unit: BG test results
Units Other Than Participants: BG test results
Arm/Group | Intended Users of the System
Number analyzed (Participants) | 115
Number analyzed (BG test results) | 115
BG test results | 115

2. Secondary Outcome: Number of Study Staff Results Within +/- 15mg/dL (<75 mg/dL) or Within +/- 20% (>=75 mg/dL) of Laboratory Glucose Method When Testing Subject Blood Glucose (BG)
Description: Study staff tested subject fingerstick blood using an investigational Blood Glucose Monitoring System (BGMS), which included an investigational meter and sensor. BGM results were compared with capillary plasma BG results obtained with a reference lab glucose method - Yellow Springs Instrument (YSI) Analyzer. BG meter results were used to calculate the number of BG results within +/- 15mg/dL (for reference BG results <75mg/dL) or +/- 20% (for reference BG results >=75mg/dL) of the reference method results.
Time Frame: 1 hour
Population: 115 (115x1) test results are possible. Staff tested blood from 118 subjects (one of 3 test strip lots). All study results from 2 subjects were excluded from data analyses as already described. Also, one test exceeded time interval (defined in protocol) between meter test and reference method.
Measure: Number; unit: BG test results
Groups:
- Study Staff: Study staff also used the investigational Blood Glucose Monitoring System (BGMS) (Tatus/Tradewind Investigational Blood Glucose Meter)
Arm/Group | Study Staff
Number analyzed (Participants) | 115
BG test results | 115

ADVERSE EVENTS:
Arm/Group | Intended Users of the System
Serious Adverse Events (participants affected / at risk) | 0/118
Other Adverse Events (participants affected / at risk) | 5/118
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intended Users of the System (N=118)
hypoglycemia (Endocrine disorders) | 5 (5) — Inclusion criteria for study stated that subjects must have diabetes. Adverse events were mild, anticipated, and not device-related.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days